CLINICAL TRIAL: NCT03831581
Title: Evaluation of Dermatomal Distribution in the Erector Spinae Plane (ESP) Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UdeA1003
Record Dates: First submitted 2019-01-14; First posted 2019-02-06 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2018-11

CONDITIONS: Pain, Chronic; Pain, Postoperative
Keywords: Erector Spinae Plane; Erector Spinae Plane Block
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Assignment interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erector Spinae Plane Block (Experimental): Patients with chest pain or upper abdomen underwent Erector Spinae Plane Block guided by ultrasound, bupivacaine 0.5% 20 ml was administered in the interfascial plane between the transverse process of T5 and the erector muscles of the spine, 60 minutes after dermatomes distribution was evaluated with pinprick and cold.
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — In patients with chest pain, ultrasound-guided Erector Spinae Plane Block block was performed at T5 transverse process in the cephalo-caudal direction with Tuohy 18 gauge needle in plane until the needle tip was located in the interfascial plane between the transverse process and the erector spinae muscles, 20 ml of bupivacaine 0.5% was administered and a catheter was inserted if indicated.

SUMMARY:
Interventional study that evaluate dermatomal distribution and its demographic determinants in patients who underwent to Erector Spinae Plane (ESP) block

DETAILED DESCRIPTION:
Interventional study that evaluate dermatomal distribution with pinprick and cold, and its demographic determinants in patients who underwent to Erector Spinae Plane (ESP) block with 20 ml of bupivacaine 0.5% at the thoracic level in patients with pain in the thorax and upper abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, in the acute / chronic pain service that presents pain in the thoracic region and / or upper hemiabdomen.

Exclusion Criteria:

* Women in pregnancy
* Patients with less than 50 Kg of weight
* Dissent of informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Dermatomes with sensitive block | 60 minutes
  Number (average) of dermatomes with sensitive block with pinprick and cold achieved at 60 minutes after the Erector Spinae Plane (ESP) block with 20 ml of bupivacaine 0.5%. Also, observe the distribution pattern.

SECONDARY OUTCOMES:
weight | 60 minutes
  weight in kilograms and its correlation with the main result The variables were grouped in means (standard deviation) for continuous variables and frequencies (percentages) for categorical variables.
Adverse events | 60 minutes and 24 hours
  Frequency of adverse events (hypotension, pneumothorax, neurological deficit, bradycardia) after the Erector Spinae Plane (ESP) block.
Success rate | 60 minutes and 24 hours
  Success rate (Blocking of at least 2 continuous dermatomes at the puncture site measured with pinprick and cold)
Degree of satisfaction | 60 minutes and 24 hours
  Degree of satisfaction evaluated with the Likert scale of 4 points (1 dissatisfied, 2 slightly dissatisfied, 3 slightly satisfied, 4 satisfied).
Visual Analogue Scale (VAS) | 60 minutes and 24 hours
  Change From Baseline in Pain Scores on the Visual analogue scale (VAS) from 1 to 10 at 60 minutes and 24 hours after the ESP block.
Height | 60 minutes
  Height in meters and its correlation with the main result The variables were grouped in means (standard deviation) for continuous variables and frequencies (percentages) for categorical variables.
Age | 60 minutes
  Age in years and its correlation with the main result The variables were grouped in means (standard deviation) for continuous variables and frequencies (percentages) for categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Cadavid, Study Chair — Universidad de Antioquia
Locations (1):
- hospital universitario San Vicente Fundacion, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No
Only final results of research

REFERENCES:
- [Derived] Barrios A, Camelo J, Gomez J, Forero M, Peng PWH, Visbal K, Cadavid A. Evaluation of Sensory Mapping of Erector Spinae Plane Block. Pain Physician. 2020 Jun;23(3):E289-E296. PMID 32517405